CLINICAL TRIAL: NCT05099744
Title: Satisfaction With Life and Quality of Life in Adults With Depressive and Anxious Symptoms: A Pilot Randomized Clinical Trial
Brief Title: Interventions in Adults With Depressive and Anxious Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Maria da Graça Pereira, Associate Professor with tenure, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EST20212022
Record Dates: First submitted 2021-09-23; First posted 2021-10-29 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; Depression
Keywords: Electrical Stimulation; Relaxation; Satisfaction with Life; Quality of Life; Psychological Morbidity
MeSH Terms: conditions — Anxiety Disorders; Depression; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized at a ratio of 1:1 for the four groups conditions. Randomization will be performed through an online random number generator by a researcher external to the team of this study, to ensure the concealment of the allocation of participants by the several groups. Only the participants will be blind to the group to which they have been allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Electrostimulation Therapy (Experimental): Participants will undergo six electrostimulation sessions, which will take place once a week and will last 20 minutes. Participants complete a set of questionnaires at the following times: pre-test (T0), post-test (T1), and 1-month post-intervention follow-up (T2). The first session will include a psychoeducational component, where it will be explained that psychological morbidity and stress influence the immune system, with repercussions on QoL.
  Interventions: Behavioral: Electrostimulation Therapy
- Relaxation + Electrostimulation Therapy (Experimental): Participants have sessions of relaxation and electrostimulation therapy during 20 minutes. They will receive two sessions in the same week, one of electrostimulation therapy and another of relaxation. Also, participants complete a set of questionnaires at the following times: pre-test (T0), post-test (T1), and 1-month post-intervention follow-up (T2).
  Interventions: Behavioral: Electrostimulation Therapy; Behavioral: Relaxation
- Relaxation (standard) (Active Comparator): Participants will receive relaxations sessions weekly, and complete a set of questionnaires at the following times: pre-test (T0), post-test (T1), and 1-month post-intervention follow-up (T2).
  Interventions: Behavioral: Relaxation
- Placebo (Placebo Comparator): Participants will be connected to the handles but will not receive any frequency during the 20 minutes. The sessions will take place at the same location and with the same weekly frequency as EG1 and EG2. Also, they will complete a set of questionnaires at the following times: pre-test (T0), post-test (T1), and 1-month post-intervention follow-up (T2).
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Electrostimulation Therapy — During 20 minutes participants are connected to the handles and receive electrostimulation therapy.
  Arms: Electrostimulation Therapy; Relaxation + Electrostimulation Therapy
Behavioral: Relaxation — During 20 minutes participants receive a session of relaxation with guided imagination. These sessions will be implemented by a trained therapist who will follow a script. The relaxation sessions are based on Schultz's autogenic relaxation training, a relaxation technique based on autosuggestion.
  Arms: Relaxation (standard); Relaxation + Electrostimulation Therapy
Behavioral: Placebo — During 20 minutes participants will be connected to the handles but will not receive any frequency.
  Arms: Placebo

SUMMARY:
In Portugal, there is an increase in cases of depression (from 6.9% to 9.8%) and anxiety (from 3.5% to 6.5%), among those enrolled in health care centers. Although the prevalence of both disorders' peaks in older adulthood, depression and anxiety often have their onset in youth. The high prevalence of psychological morbidity has been a cause for concern, given the associations between depression and anxiety in youth and other chronic mental disorders, stress, physical health problems and poorer quality of life (QoL), and physical disorders in older age.

The prevention of psychological morbidity in young people is crucial to reduce its adverse effects on young adults' development, school performance, social functioning, and to prevent its harmful impact on QoL. Cognitive behavioral therapy is considered the most effective intervention for the treatment of anxiety and depression in young people. In this study, a behavioral relaxation technique, i.e., relaxation, will be used. This technique has positive effects on psychological morbidity, specially Schultz's autogenic relaxation training.

Electrostimulation therapy, a non-invasive technique that uses electrical micro current for therapeutic purposes, is an innovative way of treating psychological morbidity, and has proven to be effective in reducing stress, depression and anxiety. Recently, studies found that cortical stimulation was associated with a reduction in depression, effects maintained after the treatment end. Also, there is evidence that there are improvements in depression, anxiety, pain and sleep, which were maintained after 4 treatment sessions.

Considering the high incidence of psychological morbidity in emerging adulthood, as well as its harmful impact on adulthood, the importance of this research aimed at reducing psychological morbidity in young adults and promoting QoL throughout life stands out. This study aims to answer the question "Does an electrostimulation therapy intervention have an impact on psychological morbidity and QoL when compared to a cognitive behavioral intervention?", with the main objective of contributing to reducing psychological morbidity in young adults, as well as promoting their QoL.

DETAILED DESCRIPTION:
The general aim of this pilot study is to assess the feasibility and acceptability of an intervention of electrostimulation versus relaxation with guided imagery (Cognitive Behavioral Therapy-TCC), according to four conditions: 1) Electrostimulation - Experimental Group 1 (EG1); 2) Relaxation with guided imagery + Electrostimulation - Experimental Group 2 (EG2); 3) Relaxation with guided imagery (standard) - Active Control Group (ACG); 4) Placebo (patients will be connected to the electrodes but receive no electrical stimulation) - Passive Control Group (PCG).

More specifically Pilot RCT specific aims:

1. Compare ACG and PCG versus EG1 and EG2, over time, on physical and psychological morbidity, emotional reactivity, perceived stress, emotional regulation, satisfaction with life and QoL.
2. To analyse the differences over time in the two experimental groups (EG1 and EG2) in physical and psychological morbidity, emotional reactivity, perceived stress, emotional regulation, life satisfaction and QoL.
3. To explore, in EG1 and EG2, the mediating role of psychological morbidity in the relationship between emotional reactivity and life satisfaction/QoL over time.
4. To explore the mediating role, in EG1 and EG2, of emotional regulation in the relationship between perceived stress, life satisfaction and QoL over time.

   The study design is longitudinal with 3 evaluation moments: pre-test (T0), post-test (T1), and 1-month post-intervention follow-up (T2). At the end of the study, the PCG will be offered the opportunity to receive intervention whether electrical stimulation or relaxation with guided imagery.

   b) Procedure The study plan is experimental (RCT) with randomization across four conditions: 1) Electrostimulation therapy - Experimental Group 1 (GE1); 2) Relaxation + Electrostimulation therapy - Experimental Group 2 (GE2); 3) Relaxation (standard) - Active Control Group (ACG); 4) Placebo (participants connected to the electrodes, but without emission of electrical frequency) - Passive Control Group (PCG).

   The young adults (students) of the different courses of the University will be contacted online for participation in the study. Participation is voluntary.

   Experimental Group (EG1 and EG2) Electrostimulation therapy will include six 20-minute sessions, weekly. The EG2 will receive two sessions in the same week, one of electrostimulation therapy and another of relaxation (CT). The first session of EG1 and EG2 will include a psychoeducational component, where it will be explained that psychological morbidity and stress influence the immune system, with repercussions on QoL, and the objective of the intervention is to reduce depressive and anxious symptoms and the impact of stress. The relaxation sessions (CT) are based on Schultz's autogenic relaxation training, a relaxation technique based on autosuggestion.

   Passive Control Group Participants in the PCG will undergo a placebo in which they will be connected to the handles but will not receive any frequency during the 20 minutes. These sessions will take place at the same location and with the same weekly frequency as EG1 and EG2.

   Active Control Group (ACG) Participants in thr ACG will undergo relaxation (CT). The sessions, as the PCG, EG1 and EG2, will have weekly frequency.

   c) Sample size calculation The sample size calculation for a pilot RCT, considering the average effect size of 0.5, a statistical power of 80% and a significance level of 5%, revealed that 12 participants were needed in each of the groups. This approach considers that one-sided 80% confidence interval for the effect size will exclude the minimum clinically significant difference if the null hypothesis is true.

   d) Data analysis To assess the feasibility of this pilot study (aim 1), the rates of eligibility, recruitment and adherence to the study protocol, participation in the follow-up and withdrawal will be calculated and its results will be presented in percentage. To obtain preliminary estimates of the intervention effects' on health outcome measures (aim 2), descriptive measures of the respective variables (means and standard deviations) will be calculated and Generalized Mixed Models will be used to check for statistically significant differences over time, in the different groups. Data will be analyzed using Statistical Package for the Social Sciences (IBM SPSS) version 27.

   e) Ethical considerations Young adults will be informed about the objectives of the study. If they accept to participate, they will be asked to complete the informed consent form. At the end of the suty, participants in the passive and active control groups will be given the opportunity to receive the relaxation intervention with guided imagination and electrostimulation therapy, respectively. The participants who, in the follow-up assessment, presented anxiety/depression symptoms above 8 will be informed of the possibility of enrolling in the Psychology Association to receive psychological support if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to present clinical levels of psychological morbidity (scores > 11 on the HADS

Exclusion Criteria:

* Personality disorder, psychosis or bipolar disorder
* Depression with psychotic features
* Suicidal ideation
* Epilepsy
* Use of defibrillator or pacemaker
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Life | Pre-test
  Satisfaction with Life it will be evaluated through Satisfaction with Life Scale with five items on a five-point Likert-Type scale, ranging from 1 "strongly disagree" to 5 "strongly agree". Scores range from 5 to 25, and higher scores suggest a greater level of satisfaction with life.
Satisfaction with Life | up to six weeks (post-test)
  Satisfaction with Life it will be evaluated through Satisfaction with Life Scale with five items on a five-point Likert-Type scale, ranging from 1 "strongly disagree" to 5 "strongly agree". Scores range from 5 to 25, and higher scores suggest a greater level of satisfaction with life.
Satisfaction with Life | 1-month post-intervention follow-up
  Satisfaction with Life it will be evaluated through Satisfaction with Life Scale with five items on a five-point Likert-Type scale, ranging from 1 "strongly disagree" to 5 "strongly agree". Scores range from 5 to 25, and higher scores suggest a greater level of satisfaction with life.
Mental and Physical Quality of Life | Pre-test
  This primary outcome it will be assessed with 12-Item Short Form Survey (SF-12). This instrument has 12 items with scores ranging from 0 to 100. Higher scores suggest a greater level of quality of life.
Mental and Physical Quality of Life | up to six weeks (post-test)
  This primary outcome it will be assessed with 12-Item Short Form Survey (SF-12). This instrument has 12 items with scores ranging from 0 to 100. Higher scores suggest a greater level of quality of life.
Mental and Physical Quality of Life | 1-month post-intervention follow-up
  This primary outcome it will be assessed with 12-Item Short Form Survey (SF-12). This instrument has 12 items with scores ranging from 0 to 100. Higher scores suggest a greater level of quality of life.

SECONDARY OUTCOMES:
Physical Morbidity | Pre-test
  This outcome it will be evaluated by the Physical Symptoms Questionnaire (PHQ-15). This instrument consists of 15 items scored on a three-point Likert-type scale ranging from 0 "not bothered at all" to 2 "bothered a lot". Scores range from 0 to 30, and higher scores indicate a greater severity of somatic symptoms.
Psychological Morbidity | up to six weeks (post-test)
  Psychological Morbidity it will be evaluated by the Hospital Anxiety and Depression Scale (HADS). This instrument has two subscales (i.e., anxiety and depression) and has 14 items scored on a four-point Likert-type scale ranging from 0 "never" to 3 "always". Scores range from 0 to 42, and higher scores indicate higher levels of anxiety and depression.
Psychological Morbidity | 1-month post-intervention follow-up
  Psychological Morbidity it will be evaluated by the Hospital Anxiety and Depression Scale (HADS). This instrument has two subscales (i.e., anxiety and depression) and has 14 items scored on a four-point Likert-type scale ranging from 0 "never" to 3 "always". Scores range from 0 to 42, and higher scores indicate higher levels of anxiety and depression.
Perceived stress | Pre-test
  This outcome it will be measured with Perceived Stress Scale (PSS). It contains 10 items rated on a five-point Likert-type scale, ranging from 0 "never" to 4 "very often". Scores range from 0 to 40, and higher scores suggest higher levels of perceived stress.
Perceived stress | up to six weeks (post-test)
  This outcome it will be measured with Perceived Stress Scale (PSS). It contains 10 items rated on a five-point Likert-type scale, ranging from 0 "never" to 4 "very often". Scores range from 0 to 40, and higher scores suggest higher levels of perceived stress.
Perceived stress | 1-month post-intervention follow-up
  This outcome it will be measured with Perceived Stress Scale (PSS). It contains 10 items rated on a five-point Likert-type scale, ranging from 0 "never" to 4 "very often". Scores range from 0 to 40, and higher scores suggest higher levels of perceived stress.
Emotional Regulation | Pre-test
  Emotional Regulation will be assessed by Difficulties in Emotion Regulation Scale (DERS). It contains 36 items on a five-point Likert-type scale ranging from 1 "rarely" applies to me" to 5 "almost always applies to me". Scores range from 36 to 180, and higher scores reflect greater impairment or dysregulation.
Emotional Regulation | up to six weeks (post-test)
  Emotional Regulation will be assessed by Difficulties in Emotion Regulation Scale (DERS). It contains 36 items on a five-point Likert-type scale ranging from 1 "rarely" applies to me" to 5 "almost always applies to me". Scores range from 36 to 180, and higher scores reflect greater impairment or dysregulation.
Emotional Regulation | 1-month post-intervention follow-up
  Emotional Regulation will be assessed by Difficulties in Emotion Regulation Scale (DERS). It contains 36 items on a five-point Likert-type scale ranging from 1 "rarely" applies to me" to 5 "almost always applies to me". Scores range from 36 to 180, and higher scores reflect greater impairment or dysregulation.
Emotional Reactivity | Pre-test
  This outcome it will be measured by Affective States Inventory-Reduced (ASI-R). This instrument is composed of a list of words that designate emotions and measure emotional states. It contains 19 items on a five-point Likert-type scale ranging from 1 "very little or not at all" to 5 "extremely". The scale contains five scales, such as negative (3 items), euphoric arousal (4 items), self-efficacy-related (4 items), Warmth (5 items) and Serenity emotions (3 items). Scores range from 3 to 15 in negative and serenity emotions subscales, from 4 to 20 in euphoric arousal and self-efficacy-related subscales, and from 5 to 25 in Warmth subscale. Higher scores indicate a higher degree to which individuals feel in the state described.
Emotional Reactivity | up to six weeks (post-test)
  This outcome it will be measured by Affective States Inventory-Reduced (ASI-R). This instrument is composed of a list of words that designate emotions and measure emotional states. It contains 19 items on a five-point Likert-type scale ranging from 1 "very little or not at all" to 5 "extremely". The scale contains five scales, such as negative (3 items), euphoric arousal (4 items), self-efficacy-related (4 items), Warmth (5 items) and Serenity emotions (3 items). Scores range from 3 to 15 in negative and serenity emotions subscales, from 4 to 20 in euphoric arousal and self-efficacy-related subscales, and from 5 to 25 in Warmth subscale. Higher scores indicate a higher degree to which individuals feel in the state described.
Emotional Reactivity | 1-month post-intervention follow-up
  This outcome it will be measured by Affective States Inventory-Reduced (ASI-R). This instrument is composed of a list of words that designate emotions and measure emotional states. It contains 19 items on a five-point Likert-type scale ranging from 1 "very little or not at all" to 5 "extremely". The scale contains five scales, such as negative (3 items), euphoric arousal (4 items), self-efficacy-related (4 items), Warmth (5 items) and Serenity emotions (3 items). Scores range from 3 to 15 in negative and serenity emotions subscales, from 4 to 20 in euphoric arousal and self-efficacy-related subscales, and from 5 to 25 in Warmth subscale. Higher scores indicate a higher degree to which individuals feel in the state described.

OTHER OUTCOMES:
Sociodemographic data | Pre-test
  The sample will be characterized using a Sociodemographic Questionnaire developed for this study (e.g., age, marital status, gender).
Clinical data | Pre-test
  The sample will be characterized using a Clinical Questionnaire developed for this study (e.g., duration of depressive and anxiety symptoms, medication).

CONTACTS AND LOCATIONS:
Overall Officials: M. Graça M. Graça Pereira, PhD, Principal Investigator — University of Minho
Locations (1):
- School of Psychology, University of Minho, Braga, Portugal

REFERENCES:
- [Background] Pandis N. Randomization. Part 3: allocation concealment and randomization implementation. Am J Orthod Dentofacial Orthop. 2012 Jan;141(1):126-8. doi: 10.1016/j.ajodo.2011.09.003. No abstract available. PMID 22196195
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Simões A. Ulterior validação de uma escala de satisfação com a vida (SWLS). Revista Portuguesa de pedagogia. 1992;26(3):503-15.
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Ferreira PL. A medição do estado de saúde: criação da versão portuguesa do MOS SF-36 [Internet]. Universidade de Coimbra, Centro de Estudos e Investigação em Saúde; 1998 [cited 2021 Sep 3]. Available from: https://estudogeral.sib.uc.pt/handle/10316/9969
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Trigo M, Canudo N, Branco F, Silva D. Estudo das propriedades psicométricas da Perceived Stress Scale (PSS) na população portuguesa. Psychologica. 2010 Dec 1;(53):353-78. doi: 10.14195/1647-8606_53_17
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment. 2004 Mar 1;26(1):41-54. doi: 10.1023/B:JOBA.0000007455.08539.94
- [Background] Coutinho J, Ribeiro E, Ferreirinha R, Dias P. Versão portuguesa da escala de dificuldades de regulação emocional e sua relação com sintomas psicopatológicos. Rev psiquiatr clín. 2010;37(4):145-51. doi: 10.1590/S0101-60832010000400001
- [Background] Moreira JM. Inventário de Estados Afetivos-Reduzido: Uma Medida Multidimensional Breve de Indicadores Emocionais de Ajustamento. 2016;14. https://www.redalyc.org/articulo.oa?id=459646901012
- [Background] Retrato da Saúde 2018 [Internet]. [cited 2021 Sep 21]. Available from: https://www.sns.gov.pt/retrato-da-saude-2018/
- [Background] Patel V, Flisher AJ, Hetrick S, McGorry P. Mental health of young people: a global public-health challenge. Lancet. 2007 Apr 14;369(9569):1302-1313. doi: 10.1016/S0140-6736(07)60368-7. PMID 17434406
- [Background] Hickey L, Hannigan A, O'Regan A, Khalil S, Meagher D, Cullen W. Psychological morbidity among young adults attending primary care: a retrospective study. Early Interv Psychiatry. 2018 Feb;12(1):22-29. doi: 10.1111/eip.12284. Epub 2015 Oct 15. PMID 26472345
- [Background] Bhattacharya R, Shen C, Sambamoorthi U. Excess risk of chronic physical conditions associated with depression and anxiety. BMC Psychiatry. 2014 Jan 16;14:10. doi: 10.1186/1471-244X-14-10. PMID 24433257
- [Background] Creswell C, Waite P, Cooper PJ. Assessment and management of anxiety disorders in children and adolescents. Arch Dis Child. 2014 Jul;99(7):674-8. doi: 10.1136/archdischild-2013-303768. Epub 2014 Mar 17. PMID 24636957
- [Background] Klainin-Yobas P, Oo WN, Suzanne Yew PY, Lau Y. Effects of relaxation interventions on depression and anxiety among older adults: a systematic review. Aging Ment Health. 2015;19(12):1043-55. doi: 10.1080/13607863.2014.997191. Epub 2015 Jan 9. PMID 25574576
- [Background] Schultz JH. Autogenic Therapy: Luthe, W. Treatment with autogenic neutralization. New York: Grune & Stratton; 1969.
- [Background] Mellen RR, Mackey W. Cranial electrotherapy stimulation (CES) and the reduction of stress symptoms in a sheriff's jail security and patrol officer population: A pilot study. American Jails. 2008;22(5):32-8.
- [Background] McClure D, Greenman SC, Koppolu SS, Varvara M, Yaseen ZS, Galynker II. A Pilot Study of Safety and Efficacy of Cranial Electrotherapy Stimulation in Treatment of Bipolar II Depression. J Nerv Ment Dis. 2015 Nov;203(11):827-35. doi: 10.1097/NMD.0000000000000378. PMID 26414234
- [Background] Bystritsky A, Kerwin L, Feusner J. A pilot study of cranial electrotherapy stimulation for generalized anxiety disorder. J Clin Psychiatry. 2008 Mar;69(3):412-7. doi: 10.4088/jcp.v69n0311. PMID 18348596
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710
- [Background] Yennurajalingam S, Kang DH, Hwu WJ, Padhye NS, Masino C, Dibaj SS, Liu DD, Williams JL, Lu Z, Bruera E. Cranial Electrotherapy Stimulation for the Management of Depression, Anxiety, Sleep Disturbance, and Pain in Patients With Advanced Cancer: A Preliminary Study. J Pain Symptom Manage. 2018 Feb;55(2):198-206. doi: 10.1016/j.jpainsymman.2017.08.027. Epub 2017 Sep 21. PMID 28870799
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344